CLINICAL TRIAL: NCT01882946
Title: A PHASE I/II CLINICAL TRIAL EVALUATING DCVax-Direct, AUTOLOGOUS ACTIVATED DENDRITIC CELLS FOR INTRATUMORAL INJECTION, IN PATIENTS WITH SOLID TUMORS
Brief Title: Safety and Efficacy Study of DCVax-Direct in Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwest Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NWBio 050012
Record Dates: First submitted 2013-06-14; First posted 2013-06-21 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Locally Advanced Tumor; Metastatic Solid Tissue Tumors; Liver Cancer; Colorectal Cancer; Pancreatic Cancer; Melanoma
MeSH Terms: conditions — Liver Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DCVax-Direct (Experimental): DCVax-Direct: autologous, activated dendritic cells for intratumoral injection
  Interventions: Biological: DCVax-Direct

INTERVENTIONS:
Biological: DCVax-Direct — Autologous, activated dendritic cells for intratumoral injection

SUMMARY:
The study comprises a Phase I component during which the optimal dose of DCVax-Direct for the treatment of solid tissue tumors will be identified, followed by a Phase II component to determine if the injection of DCVax-Direct into selected solid tissue tumors has the ability to reduce tumor growth.

ELIGIBILITY:
Inclusion Criteria (summary):

* Age between 18 and 75 years (inclusive) at screening.
* Karnofsky performance status (KPS) of 70 or higher or Eastern Cooperative Oncology Group (ECOG) 0-1 at screening.
* Subjects with a histological or cytopathological confirmed diagnosis of a locally advanced or metastatic solid tumor malignancy for which primary treatment is no longer effective or does not offer curative or life-prolonging potential per clinician judgment, with the understanding that DCVax-Direct is not intended as a treatment of last resort.
* Not eligible for complete resection due to either tumor location, physician's assessment or subject's choice.
* Must have completed at least one recent treatment regimen in the metastatic or advanced setting in the disease currently under treatment to reduce tumor burden.
* Any steroid therapy >2 mg dexamethasone or equivalent dose should be stopped or have been tapered down 2 weeks prior to the leukapheresis.
* At least one measurable tumor mass, i.e. a lesion that can accurately be measured by CT/MRI in at least one dimension with longest diameter ≥ 1 cm, that is accessible for injection either with or without imaging (CT/ultrasound) guidance.
* Adequate hematological, hepatic, and renal function,
* Adequate blood coagulation parameters
* Life expectation of >3 months.

Exclusion Criteria (Summary):

* Positive HIV-1, HIV-2, or Human T-lymphotropic virus (HTLV-I/II) tests.
* History of current or prior (within the last two years) active clinically significant malignancy other than the tumor type for which DCVax-Direct treatment is considered, and except for primary tumor in the case of metastases and adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Heavily pretreated (HP) subjects are not eligible for this study, unless treatments have occurred more than 1 year in the past.
* Presence of brain metastases, unless treated surgically and/or irradiated and clinically stable off steroids or on low dose (< 2 mg per day) steroids for ≥ 14 days, or presence of leptomeningeal disease.
* History of immunodeficiency or unresolved autoimmune disease.
* Requirement for ongoing immunosuppressants.
* Prior active immunotherapy for cancer within the past 2 years.
* Ongoing medical need for continuous anti-coagulation or anti-platelet medication.
* Known genetic cancer-susceptibility syndromes.
* Acute or active uncontrolled infection
* Ongoing fever ≥ 101.5 degrees F/38.6 degrees C at screening.
* Unstable or severe intercurrent medical conditions such as unstable angina, uncontrolled arrhythmias, Crohn's Disease, ulcerative colitis etc.
* Females of child-bearing potential who are pregnant or lactating or who are not using adequate contraception (surgical, hormonal or double barrier, i.e. condom and diaphragm).
* Allergy or anaphylaxis to any of the reagents used in this study.
* Inability to obtain informed consent because of psychiatric or complicating medical problems.
* Inability or unwillingness to return for required visits and follow-up exams.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | 6 months

SECONDARY OUTCOMES:
Number of patients with tumor response | 18 months

OTHER OUTCOMES:
Number of patients surviving | 24 months
Number of patients surviving without tumor progression | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Marnix Bosch, MBA, PhD, Study Director — Northwest Biotherapeutics
Locations (2):
- United States (2):
  - Orlando Health, Orlando, Florida
  - MD Anderson Cancer Center, Houston, Texas